CLINICAL TRIAL: NCT02897921
Title: Clinical Importance of Carrier Status of Recessive Gene Mutations in Myopathy
Brief Title: Clinical Importance of Carrier Status of Recessive Gene Mutations in Myopathy (CICS)
Acronym: CICS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tove Freja Maria Fornander, Student researcher, Rigshospitalet, Denmark
Other Study IDs: H-16035677
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Recessive Gene Myopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Carriers of recessive gene mutations of myopathies: Patients with several different kinds of recessively inherited myopathy genes, such as for example Duchenne's Muscular Dystrophy, Becker's Muscular Dystrophy, Limb Girdle limb girdle muscle dystrophy (LGMD) type 2A and 2L etc.
  Investigated by blood sampling, Biodex 4 Isokinetic Dynamometer, MRI analysis, ECG, Holter monitoring, and echocardiography.
- Healthy controls: Healthy controls, investigated by blood sampling, Biodex 4 Isokinetic Dynamometer and MRI analysis.

SUMMARY:
Many myopathies are inherited in a recessive manner, but in some of these recessively inherited disorders, clinical manifestations may potentially manifest in carriers of just a single mutation.

The aim of the study is to describe the clinical characteristics of single mutation carriers of recessive myopathy, through measuring serum creatine kinase, muscle strength, muscle degeneration (by MRI) and heart affection. The investigators will do this by blood sampling, Biodex 4 Isokinetic Dynamometer, MRI analysis, ECG, Holter monitoring, and echocardiography.

The aim is further to describe whether these characteristics are found primarily with specific mutations.

DETAILED DESCRIPTION:
Background:

Many myopathies are inherited in a recessive manner, but in some of these recessively inherited disorders, clinical manifestations may potentially manifest in carriers of just a single mutation. This has recently been demonstrated by researchers for the recessively inherited limb girdle muscle dystrophy (LGMD) type 2A, where carriers of single mutations can also be symptomatic. In X-linked recessively inherited dystrophinopathies caused by mutations in the DMD gene on chromosome Xp21, female mutation carriers may also manifest with disease, although this is often milder than affected men. In the recently discovered LGMD2L, manifesting carriers are also suspected. Thus, according to statistics, too many persons evaluated for myopathy carry a single LGMD2L mutation.

Some previous studies have looked into the significance of being a single mutation carrier in recessive muscle disease. In dystrophinopathy, it was reported that 5 % of female DMD carriers reported myalgia and cramps, 17 % experienced mild-to-moderate muscle weakness and 8 % experienced dilated cardiomyopathy, with a mean onset age of approximately 30 years. Another study found that echocardiographic examination was abnormal in up to 38% of DMD female carriers - some with dilated cardiomyopathy, and some with left ventricle dilatation.

Overall, however significance of carrying a single mutation of recessive myopathy is widely unexplored. No study has yet investigated the characteristics of single mutation carriers of recessive myopathy in an observational, cross-sectional study.

Aim:

In this study, clinical characteristics of single mutation carriers of recessive myopathies will be investigated. The investigation will include sceletal muscle degeneration and strength, as well as cardiac status.

Recruitment and Methods:

Estimated total of subjects recruited is 200 with known recessive gene mutations, and 40 healthy controls. In former studies 40 healthy volunteers have already been investigated, thereby giving a total of 80 healthy controls. Recessive gene carrier recruits will be obtained via the Department of Clinical Genetics and Copenhagen Neuromuscular Center, Rigshospitalet, thus only including carriers aware of their carrier status.

2 days of testing per participant. Day one: Measuring S-creatine kinase level (blood sampling), muscle strength (Biodex 4 Isokinetic Dynamometer), ECG, and Holter monitor device application.

Day two: Holter monitor device removal, Dixon MRI analysis with gadolinium contrast medium, and echocardiography.

Healthy controls will take part in MRI-scanning and isokinetic dynamometer testing.

Trials are expected to be carried out between October 2016 and May 2020.

ELIGIBILITY:
Single mutation carriers of recessive myopathy:

Inclusion Criteria:

* Verified carrier status of recessive myopathy mutation before entry into the study
* Age of 18 years or older

Exclusion Criteria:

* Contraindications for MRI (pacemaker or other internal metal or magnetic devices)
* Claustrophobia
* Pregnancy at the time of MRI
* After investigators judgement

Healthy controls:

Inclusion Criteria:

• Age of 18 years or older

Exclusion Criteria:

* Contraindications for MRI (pacemaker or other internal metal or magnetic devices)
* Claustrophobia
* Pregnancy at the time of MRI
* After investigators judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2 groups are studied: 1) Single mutation carriers of recessive myopathies. 2) Healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Cardiac status | MRI of cardiac status and muscles takes around 1,5 hours
  We will use MRI with a contrast agent (gadolinium). Kidney function and contrast allergy status will be tested prior to use of contrast agent, and avoided if the participant is not suitable for contrast injection.
Muscle tissue quality | MRI of cardiac status and muscles takes around 1,5 hours
  Muscle tissue cross sectional area and fat percent will be investigated and measured by Dixon MRI scan.

SECONDARY OUTCOMES:
Serum CK-levels | Estimated time 5 minutes.
  Blood sampling
Muscle strength | Testing takes around 10-20 minutes
  Investigated by an isokinetic dynamometer (Biodex 4).
ECG | Estimated time: 5 minutes.
  ECG electrodes will be places on the subject's chest, and an electrocardigram will be measured.
Holter monitor | A Holter monitor device will be attached on test day 1, and worn until test day 2 (24-48 hours)
  The electrodes will be places on the chest and the monitor attached in a line around the neck. 24-48 hours of electrocardiogram will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Tove Freja M Fornander, B. Sc., Principal Investigator — Copenhagen Neuromuscular Center
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet, 3342, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Hoogerwaard EM, van der Wouw PA, Wilde AA, Bakker E, Ippel PF, Oosterwijk JC, Majoor-Krakauer DF, van Essen AJ, Leschot NJ, de Visser M. Cardiac involvement in carriers of Duchenne and Becker muscular dystrophy. Neuromuscul Disord. 1999 Jul;9(5):347-51. doi: 10.1016/s0960-8966(99)00018-8. PMID 10407858
- [Background] Lee SH, Lee JH, Lee KA, Choi YC. Clinical and Genetic Characterization of Female Dystrophinopathy. J Clin Neurol. 2015 Jul;11(3):248-51. doi: 10.3988/jcn.2015.11.3.248. Epub 2015 May 28. PMID 26022459
- [Background] Vissing J, Barresi R, Witting N, Van Ghelue M, Gammelgaard L, Bindoff LA, Straub V, Lochmuller H, Hudson J, Wahl CM, Arnardottir S, Dahlbom K, Jonsrud C, Duno M. A heterozygous 21-bp deletion in CAPN3 causes dominantly inherited limb girdle muscular dystrophy. Brain. 2016 Aug;139(Pt 8):2154-63. doi: 10.1093/brain/aww133. Epub 2016 Jun 3. PMID 27259757
- [Background] Flanigan KM. Oxford Textbook of Neuromuscular Disorders chapter 22 "The dystrophinopathies". Oxford University Press 2014, first edition.